CLINICAL TRIAL: NCT03308721
Title: A Multiple Dose Trial Investigating Safety, Tolerability and Pharmacokinetics for Multiple Doses of NNC9204-1177 in Subjects Being Overweight or With Obesity
Brief Title: Research Study Investigating Study Medicine (NNC9204-1177) for Weight Management in People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9277-4328; U1111-1189-1919 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC9204-1177 (Experimental): Dose trial with a sequential trial design
  Interventions: Drug: NNC9204-1177 A 1.0 mg/mL
- Placebo (Placebo Comparator)
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: NNC9204-1177 A 1.0 mg/mL — Participants will get 1 or more injections into the skin of the stomach area once each week for 12 weeks.
  Dose gradually increased to 6000 μg.
  Arms: NNC9204-1177
Drug: PLACEBO — Participants will get 1 or more injections into the skin of the stomach area once each week for 12 weeks.
  Arms: Placebo

SUMMARY:
This study looks at a new study medicine for weight management in people with overweight or obesity. The aim of this study is to find out how safe and tolerable the study medicine is. The study also looks at how the study medicine behaves in the body and how it is removed from the body.

Participants will either get NNC9204-1177 (the new study medicine) or placebo (a formula that looks like the study medicine but does not have active ingredients). Which treatment participants get will be decided by chance.

NNC9204-1177 has not been approved by the United States Food and Drug Administration. Its use in this study is experimental. Participants will get 1 or more injections into the skin of the stomach area once each week for 12 weeks.

The study will last for about 5 months. Participants will have 19 clinic visits with the study doctor. At certain times during the study, participants will have blood draws and 3 different kinds of electrocardiograms. Participants will answer mental health questionnaires. Women: Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 27.0 and 39.9 kg/m2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol
* Subjects, aged at least 40 years, with an estimated 10-year atherosclerotic cardiovascular disease (ASCVD) risk greater than or equal to 5%
* Male subjects who are not sexually abstinent or surgically sterilised (vasectomy) and are sexually active with female partner(s) who are not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their non-pregnant female partner(s) (Pearl Index below 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide), or who intend to donate sperm in the period from screening until 3 months following last administration of the investigational medical product
* Female subjects who are of child bearing potential (pre-menopausal and not surgically sterilised) and are sexually active with male partner(s) who are not surgically sterilised (vasectomy) and who are not using highly effective contraceptive methods (Pearl Index below 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide) combined with a highly effective method of contraception for their male partner(s) (e.g. condom with spermicide), or who are pregnant, breast-feeding or intend to become pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | Day 1-110
  Count of events

SECONDARY OUTCOMES:
The area under the NNC9204-1177 serum concentration-time curve at steady state | 0-168 hours
  Calculated based on NNC9204-1177 measured in blood.
The maximum serum concentration of NNC9204-1177 at steady state | Day 78-110
  Calculated based on NNC9204-1177 measured in blood.
The time to maximum serum concentration of NNC9204-1177 | Day 78-110
  Calculated based on NNC9204-1177 measured in blood.
The terminal half-life of NNC9204-1177 from steady state | Day 78-110
  Calculated based on NNC9204-1177 measured in blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Skovgaard D, Haahr PM, Lester R, Clark K, Paglialunga S, Finer N, Friedrichsen MH, Hjerpsted JB, Engelmann MDM. Prevalence of Baseline Cardiac Arrhythmias in Participants with Overweight or Obesity in Phase 1 Clinical Trials: Analysis of 24-Hour Holter Electrocardiogram Recordings. J Clin Pharmacol. 2023 May;63(5):539-543. doi: 10.1002/jcph.2193. Epub 2023 Jan 20. PMID 36524539